CLINICAL TRIAL: NCT00006449
Title: Post-Treatment Effects of Naltrexone
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: NIAAADAV12696; R01AA012696 (NIH)
Record Dates: First submitted 2000-11-06; First posted 2000-11-07 (Estimated); Last update posted 2010-05-12 (Estimated); Status verified 2010-05

CONDITIONS: Alcoholism
MeSH Terms: conditions — Alcoholism | interventions — Naltrexone; Motivational Interviewing

INTERVENTIONS:
Drug: naltrexone (Revia)
Behavioral: broad spectrum treatment
Behavioral: motivational enhancement therapy

SUMMARY:
The aims of this protocol are to compare 3 and 6 months of naltrexone treatment coupled with two psychotherapies that differ in scope and intensity. The effect of these treatments will be assessed with patients who differ in their psychosocial need and resources at their disposal, and in their level of cravings for alcohol.

ELIGIBILITY:
Inclusion Criteria:

* Meets current diagnosis of alcohol dependence and have been abstinent for a minimum of 3 and maximum of 21 days prior to treatment
* Must be able to participate in an 18-month outpatient study, and live within a one hour or less commute to treatment facility.
* Must be fluent in English.
* Women of childbearing potential must have a negative pregnancy test.

Exclusion Criteria:

* Severe hepatic disease or a liver function test greater than 4 times normal.
* Opiate use in the last 14 days or a history of opioid dependence in the past year.
* Pregnant or lactating females who are not using a reliable method of birth control.
* Inability to follow medication instructions and safety precautions.
* Comorbid substance dependence diagnosis in the past 6-months, excluding nicotine or marijuana dependence.
* Use of medications intended to decrease drinking.
* Meets criteria for bipolar disorder, schizophrenia, bulimia/anorexia, dementia, major depression.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160
Dates: Start 2000-09; Study Completion 2006-07

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Psychiatric Research, Indiana University School of Medicine, Indianapolis, Indiana, United States